CLINICAL TRIAL: NCT02963974
Title: Cochlear Implantation in Pediatric Cases of Unilateral Hearing Loss
Acronym: CIPUHL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Med-El Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-3350
Record Dates: First submitted 2016-10-27; First posted 2016-11-15 (Estimated); Results first posted 2021-08-05 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-06

CONDITIONS: Hearing Loss, Unilateral
Keywords: cochlear implant
MeSH Terms: conditions — Hearing Loss, Unilateral | interventions — Cochlear Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Cochlear Implant (Experimental): Pediatric patients with single sided deafness will receive a cochlear implant in the ear of loss
  Interventions: Device: Cochlear implant

INTERVENTIONS:
Device: Cochlear implant — Implantation
  Other Names: MED-EL Cochlear Implant; MED-EL Synchrony with FLEX 28 array; MED-EL Synchrony with FLEX 24 array

SUMMARY:
This feasibility study evaluates whether children with unilateral, moderate to profound sensorineural hearing loss experience an improvement in speech perception, hearing in noise, localization, and quality of life with a cochlear implant as compared to an unaided listening condition.

DETAILED DESCRIPTION:
Unilateral hearing loss (UHL) is a term used to describe a substantial hearing loss in one ear and normal hearing in the contralateral ear. Despite normal hearing in one ear, these individuals experience reduced speech perception in noise, variable abilities on localization tasks, increased reports of hearing handicap, reduced quality of life, and often, they obtain limited or no benefit from conventional amplification. In the United States, the prevalence of UHL in children ranges from 0.03% to 3%, depending on the age of the child.

Cochlear implantation performed for children with bilateral, severe to profound deafness has significant impacts on several aspects of child development.

The practice of providing cochlear implants to children who have significant hearing loss in one ear is of great interest and is occurring with greater frequency as reported in case studies and small set clinical reports. The primary purpose of this feasibility study is to demonstrate the effectiveness of cochlear implantation in children, age 3 years 6 months to 6 years, 6 months, with moderate to profound UHL. Postoperative results will be evaluated with speech perception measures, localization tasks, hearing in noise tasks, and subjective reports.

ELIGIBILITY:
i) Inclusion Criteria

1. Unilateral moderate-to-profound sensorineural hearing loss.

   1. Unaided residual hearing thresholds that yield a pure tone average (PTA) at frequencies 500 Hz, 1 kHz and 2 kHz of ≥70 dB HL in the ear to be implanted. It is possible that subjects may have hearing at other frequencies not included in this average.
   2. Hearing thresholds in the contralateral ear of ≤25 dB HL
2. Between 3 years, 6 mos and 6 years, 6 mos of age at implantation.
3. Anatomically normal cochlear nerve
4. Cochlear anatomy that is amenable to cochlear implantation as evaluated by imaging (modality at the physician's discretion) including:

   1. Normal cochlear anatomy or
   2. Incomplete Partition Type II (IP2) with or without Enlarged Vestibular Aqueduct (EVA) or
   3. EVA with normal partitioning
5. No evidence of progressive hearing loss.
6. Willing to undergo 4 week hearing aid trial as warranted based on achieving desired audibility when fitted via real ear desired sensation level (DSL) method.
7. Aided word recognition in the ear to be implanted of 30% or less as measured with Consonant Nucleus Consonant (CNC) words (50-word list)

   1. When listening with an appropriately fit hearing aid and masking applied to the contralateral ear (Turner, 2004).
   2. Aided testing will be conducted in a sound-proof booth with the participant seated 1 meter from the sound source, facing 0° azimuth. Recorded materials will be presented at 60 dB SPL.
   3. The hearing aid output will be measured using DSL targets.
8. Realistic parental expectations: a verbal acknowledgement of the potential benefits and risks, and postoperative variation in performance. For instance, cochlear implantation will not restore normal hearing.
9. Willing to obtain recommended meningitis vaccinations per CDC recommendations.

(9) Development and cognition within the normal range as measured by the Leiter-R test of nonverbal intelligence and cognitive abilities and the Bracken Basic Concept Scale -Revised.

(10) Parental commitment to study parameters including being able and willing to participate in evaluation schedule, involvement in prescribed therapy, and travel to investigational site and study-related activities.

ii) Exclusion Criteria

1. English is not primary language of the home

   1. Speech perception materials are presented in English
   2. Parental questionnaires are administered in English
2. Conductive hearing loss in either ear
3. Compromised auditory nerve
4. Ossification of the cochlea
5. Inability to participate in follow-up procedures (i.e., unwillingness, geographic location)
6. History of condition that contraindicates middle or inner ear surgery or anesthesia (i.e. otitis media refractory to treatment)
7. Case of sudden sensorineural hearing loss that has not been first evaluated by a physician

Ages: 42 Months to 78 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2021-05-07 (Actual); Study Completion 2021-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin D Brown, MD, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arndt S, Aschendorff A, Laszig R, Beck R, Schild C, Kroeger S, Ihorst G, Wesarg T. Comparison of pseudobinaural hearing to real binaural hearing rehabilitation after cochlear implantation in patients with unilateral deafness and tinnitus. Otol Neurotol. 2011 Jan;32(1):39-47. doi: 10.1097/MAO.0b013e3181fcf271. PMID 21068690
- [Background] Firszt JB, Holden LK, Reeder RM, Waltzman SB, Arndt S. Auditory abilities after cochlear implantation in adults with unilateral deafness: a pilot study. Otol Neurotol. 2012 Oct;33(8):1339-46. doi: 10.1097/MAO.0b013e318268d52d. PMID 22935813
- [Background] Bess FH, Tharpe AM, Gibler AM. Auditory performance of children with unilateral sensorineural hearing loss. Ear Hear. 1986 Feb;7(1):20-6. doi: 10.1097/00003446-198602000-00005. PMID 3949097
- [Background] Arndt S, Prosse S, Laszig R, Wesarg T, Aschendorff A, Hassepass F. Cochlear implantation in children with single-sided deafness: does aetiology and duration of deafness matter? Audiol Neurootol. 2015;20 Suppl 1:21-30. doi: 10.1159/000380744. Epub 2015 May 19. PMID 25999052
- [Background] Kompis M, Pfiffner F, Krebs M, Caversaccio MD. Factors influencing the decision for Baha in unilateral deafness: the Bern benefit in single-sided deafness questionnaire. Adv Otorhinolaryngol. 2011;71:103-111. doi: 10.1159/000323591. Epub 2011 Mar 8. PMID 21389710
- [Background] Varni JW, Limbers CA, Burwinkle TM. Impaired health-related quality of life in children and adolescents with chronic conditions: a comparative analysis of 10 disease clusters and 33 disease categories/severities utilizing the PedsQL 4.0 Generic Core Scales. Health Qual Life Outcomes. 2007 Jul 16;5:43. doi: 10.1186/1477-7525-5-43. PMID 17634123
- [Background] PETERSON GE, LEHISTE I. Revised CNC lists for auditory tests. J Speech Hear Disord. 1962 Feb;27:62-70. doi: 10.1044/jshd.2701.62. No abstract available. PMID 14485785
- [Background] Galvin KL, Noble W. Adaptation of the speech, spatial, and qualities of hearing scale for use with children, parents, and teachers. Cochlear Implants Int. 2013 Jun;14(3):135-41. doi: 10.1179/1754762812Y.0000000014. PMID 23394704
- [Derived] Park LR, Dillon MT, Buss E, Brown KD. Two-Year Outcomes of Cochlear Implant Use for Children With Unilateral Hearing Loss: Benefits and Comparison to Children With Normal Hearing. Ear Hear. 2023 Sep-Oct 01;44(5):955-968. doi: 10.1097/AUD.0000000000001353. Epub 2023 Mar 7. PMID 36879386

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cochlear Implant
Started | 20
Completed | 19
Not Completed | 1

BASELINE CHARACTERISTICS:
Population: Ethnicity data were not collected,
Arm/Group | Cochlear Implant
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.5 (2.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 14
  More than one race | 3
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20
Ear Affected [Count of Participants; unit: Participants]
  Left Ear | 10
  Right Ear | 10
Etiology of Hearing Loss [Count of Participants; unit: Participants]
  Unknown | 12
  Congenital Cytomegalovirus | 3
  Mondini Malformation | 2
  Infection | 1
  Trauma | 1
  Waardenburg Syndrome | 1
Suspected Length of Deafness [Mean (Standard Deviation); unit: years] | 3.3 (1.7)

OUTCOME MEASURES:

1. Primary Outcome: Change Over Time in the Ability to Perceive Single Words as Assessed by Consonant-Nucleus-Consonant (CNC) Word Recognition Testing
Description: Recorded, open set word recognition presented pre-operatively in the soundfield when using a traditional hearing aid (contralateral ear masked) and at 3-, 6-, 9-, 12-, 18-, and 24-month post-activation intervals by direct input to the speech processor using the Consonant-Nucleus-Consonant (CNC) words. Scores are reported as percent words correct and a higher score is better. Change is measured from the pre-operative to the 3-month post-activation interval, and from the 3-month post-activation interval to each subsequent interval.
Time Frame: up to 24 months post-activation
Population: One participant was lost to follow-up after Month 12
Measure: Mean (Standard Deviation); unit: percentage of words correct
Arm/Group | Cochlear Implant
Number analyzed (Participants) | 20
percentage of words correct
  Pre-operatively | 1.4 (6.3)
  Month 3 | 14.4 (14.5)
  Month 6 | 28.2 (18.0)
  Month 9 | 45.0 (15.2)
  Month 12 | 50.3 (33.1)
  Month 18: number analyzed (Participants) | 19
  Month 18 | 51.8 (11.3)
  Month 24: number analyzed (Participants) | 19
  Month 24 | 58.6 (15.4)
Statistical Analysis 1: Comparison: Cochlear Implant; Analyzed CNC Word scores from 3 months through 24 months to evaluate change over time with device use. Scores were converted to Rau prior to analysis; Test type: Superiority; p < 0.001, Mixed Models Analysis — The a priori threshold for statistical significance was < 0.05
Statistical Analysis 2: Comparison: Cochlear Implant; Analyzed pre-op to 3 month post activation CNC Word scores to test superiority of cochlear implant use to pre-operative hearing aid use; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney) — The a priori threshold for statistical significance was p < 0.05

2. Primary Outcome: Mean Change in the Signal-to-noise Ratio 50 (SNR-50) From Device Off to Device on as Measured With the Bamford-Kowal-Bench Speech in Noise Test (BKB-SIN) at 6 Months Post-activation
Description: Two ½ lists of the BKB-SIN were presented in each condition device off and device on after 6-months of device use: Speech and masker in front, speech in front and masker directed 90 degrees to the normal ear, speech in front and masker directed 90 degrees to the affected ear. The SNR-50 represents the signal-to-noise ratio required to perceive 50% of the sentence. A lower score is better.
Time Frame: 6 months post-activation
Measure: Mean (95% Confidence Interval); unit: signal-to-noise ratio
Arm/Group | Cochlear Implant
Number analyzed (Participants) | 20
signal-to-noise ratio
  Device off to device on with speech and noise in front | 1.8 [0.4 to 3.2]
  Device off to device on with speech in front and noise to the implanted side | 0.4 [-1.2 to 1.9]
  Device off to device on with speech in front and noise to the normal side | 1.9 [0.4 to 3.5]

3. Primary Outcome: Mean Change in the SNR-50 From Device Off to Device on as Measured With the BKB-SIN at 12 Months Post-activation
Description: Two ½ lists of the BKB-SIN were presented in each condition device off and device on after 12-months of device use: Speech and masker in front, speech in front and masker directed 90 degrees to the normal ear, speech in front and masker directed 90 degrees to the affected ear. The SNR-50 represents the signal-to-noise ratio required to perceive 50% of the sentence. A lower score is better.
Time Frame: 12 months post-activation
Measure: Mean (95% Confidence Interval); unit: signal-to-noise ratio
Arm/Group | Cochlear Implant
Number analyzed (Participants) | 20
signal-to-noise ratio
  Device on with speech and noise in front | 1.6 [0.5 to 2.7]
  Device off to device on with speech in front and noise to the implanted side | 2.5 [1.1 to 3.9]
  Device off to device on with speech in front and noise to the normal side | 3.5 [1.8 to 5.2]
Statistical Analysis 1: Comparison: Cochlear Implant; Analyzed BKB-SIN SNR-50 scores at 12 months post activation to evaluate the impact of device use (CI off vs on) and masker location (front, to the affected ear, or to the normal hearing ear) on hearing in noise; Test type: Superiority; p < 0.001, ANOVA — The a priori threshold for statistical significance was < 0.05. This was a two-way repeated measures ANOVA

4. Primary Outcome: Mean Change in the SNR-50 From Device Off to Device on as Measured With the BKB-SIN at 24 Months of Device Use
Description: Two ½ lists of the BKB-SIN were presented in each condition device off and device on after 24-months of device use: Speech and masker in front, speech in front and masker directed 90 degrees to the normal ear, speech in front and masker directed 90 degrees to the affected ear. The SNR-50 represents the signal-to-noise ratio required to perceive 50% of the sentence. A lower score is better.
Time Frame: 24 months post-activation
Population: One participant was lost to follow-up after Month 12
Measure: Mean (95% Confidence Interval); unit: signal-to-noise ratio
Arm/Group | Cochlear Implant
Number analyzed (Participants) | 19
signal-to-noise ratio
  Device off to device on with speech and noise in front | 1.4 [-0.1 to 2.8]
  Device off to device on with speech in front and noise to the implanted side | 1.7 [0.0 to 3.4]
  Device off to device on with speech in front and noise to the normal side | 4.0 [2.6 to 5.4]
Statistical Analysis 1: Comparison: Cochlear Implant; Analyzed BKB-SIN SNR-50 scores across all time points (6, 12, and 24 months post activation) to evaluate the impact of time, device use (CI off vs on), and masker location (front, to the affected ear, or to the normal hearing ear) on hearing in noise; Test type: Superiority; p < 0.001, Mixed Models Analysis — The a priori threshold for statistical significance was < 0.05

5. Primary Outcome: Median Change in Localization Error From Device Off to Device on at 3 Months Post-activation
Description: Soundfield localization of 200-ms speech-shaped noise, presented from 11 speakers at 70 decibel (dB) sound pressure level (SPL) in a sound treated room. Error measures are made device on and device off after 3 months of device use. Overall root-mean-square (RMS) error is the difference between the sound source azimuth and the response azimuth and a lower score indicates more accurate localization of the sound source. Random error is the average of the standard deviation of the responses for each source and a lower score reflects a more consistently accurate response. Constant error is a measure of side bias, and a lower score indicates less response bias to either side. Adjusted constant error is a measure of reliability in the response taking side bias into account, and a lower score indicates a more reliable response.
Time Frame: 3 months post-activation
Measure: Median (95% Confidence Interval); unit: degrees
Arm/Group | Cochlear Implant
Number analyzed (Participants) | 20
degrees
  Overall RMS error from device off to device on | 14.7 [3.5 to 31.8]
  Random error from device off to device on | -0.8 [-5.1 to 9.3]
  Constant error from device off to device on | 18.8 [4.0 to 32.2]
  Adjusted constant error from device off to device on | 19.1 [3.0 to 26.0]

6. Primary Outcome: Median Change in Localization Error From Device Off to Device on at 9 Months Post-activation
Description: Soundfield localization of 200-ms speech-shaped noise, presented from 11 speakers at 70 decibel (dB) sound pressure level (SPL) in a sound treated room. Error measures are made device on and device off after 9 months of device use. Overall root-mean-square (RMS) error is the difference between the sound source azimuth and the response azimuth and a lower score indicates more accurate localization of the sound source. Random error is the average of the standard deviation of the responses for each source and a lower score reflects a more consistently accurate response. Constant error is a measure of side bias, and a lower score indicates less response bias to either side. Adjusted constant error is a measure of reliability in the response taking side bias into account, and a lower score indicates a more reliable response.
Time Frame: 9 months post-activation
Measure: Median (95% Confidence Interval); unit: degrees
Arm/Group | Cochlear Implant
Number analyzed (Participants) | 20
degrees
  Overall RMS error from device off to device on | 24.6 [16.9 to 28.2]
  Random error from device off to device on | 15.8 [8.2 to 18.5]
  Constant error from device off to device on | 27.9 [8.3 to 35.1]
  Adjusted constant error from device off to device on | 24.9 [7.6 to 33.0]

7. Primary Outcome: Median Change in Localization RMS Error From Device Off to Device on at 18 Months Post-activation
Description: Soundfield localization of 200-ms speech-shaped noise, presented from 11 speakers at 70 decibel (dB) sound pressure level (SPL) in a sound treated room. Error measures are made device on and device off after 18 months of device use. Overall root-mean-square (RMS) error is the difference between the sound source azimuth and the response azimuth and a lower score indicates more accurate localization of the sound source. Random error is the average of the standard deviation of the responses for each source and a lower score reflects a more consistently accurate response. Constant error is a measure of side bias, and a lower score indicates less response bias to either side. Adjusted constant error is a measure of reliability in the response taking side bias into account, and a lower score indicates a more reliable response.
Time Frame: 18 months post-activation
Population: One participant was lost to follow-up after Month 12
Measure: Median (95% Confidence Interval); unit: degrees
Arm/Group | Cochlear Implant
Number analyzed (Participants) | 19
degrees
  RMS error from device off to device on | 37.7 [18.0 to 50.5]
  Random error from device off to device on | 20.2 [11.2 to 24.6]
  Constant error from device off to device on | 27.5 [15.6 to 46.9]
  Adjusted constant error from device off to device on | 24.9 [11.4 to 39.1]

8. Primary Outcome: Median Change in Localization Error From Device Off to Device on at 24 Months Post-activation
Description: Soundfield localization of 200-ms speech-shaped noise, presented from 11 speakers at 70 decibel (dB) sound pressure level (SPL) in a sound treated room. Error measures are made device on and device off after 24 months of device use. Overall root-mean-square (RMS) error is the difference between the sound source azimuth and the response azimuth and a lower score indicates more accurate localization of the sound source. Random error is the average of the standard deviation of the responses for each source and a lower score reflects a more consistently accurate response. Constant error is a measure of side bias, and a lower score indicates less response bias to either side. Adjusted constant error is a measure of reliability in the response taking side bias into account, and a lower score indicates a more reliable response.
Time Frame: 24 months post-activation
Population: One participant was lost to follow-up after Month 12
Measure: Median (95% Confidence Interval); unit: degrees
Arm/Group | Cochlear Implant
Number analyzed (Participants) | 19
degrees
  RMS error from device off to device on | 35.1 [15.1 to 47.0]
  Random error from device off to device on | 17.9 [7.6 to 28.4]
  Constant error from device off to device on | 25.8 [9.3 to 39.3]
  Adjusted constant error from device off to device on | 21.1 [8.9 to 39.9]
Statistical Analysis 1: Comparison: Cochlear Implant; Analyzed overall RMS error at 3, 9, 18, and 24 months post activation to evaluate the impact of device use (CI off vs on) and time on localization; Test type: Superiority; p = 0.01911, Mixed Models Analysis — The a priori threshold for statistical significance was < 0.05

9. Primary Outcome: Change in Mean Response Scores on the Speech Spatial & Qualities (SSQ) Questionnaire
Description: The Speech Spatial Qualities Questionnaire requires participants to rate their perceived hearing ability for 49 scenarios using a 10-point scale, ranging from 0 (Not at all) to 10 (Perfectly). A score higher than 0 for each listening scenario shows some benefit of the device, while a score of 10 indicates the device was extremely beneficial. The SSQ questionnaire assesses performance in 3 domains, hearing speech in quiet and noise environments (9 items), spatial or directional hearing (5 items) and sound qualities (8 items). Domain scores represent an average of item ratings, therefore each domain score ranges from 0 to 10 with a higher score indicating a better outcome. The pediatric version of this test was used and parents reported as proxy pre-operatively and at at 3-, 6-, 9-, 12-, 18-, and 24-month post-activation intervals. Change is measured from the pre-operative to the 3-month post-activation interval and between the 3-month interval to all subsequent intervals.
Time Frame: Pre-operatively through 24 months post-activation
Population: One participant was lost to follow-up after Month 12
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Cochlear Implant
Number analyzed (Participants) | 20
score on a scale
  Speech: pre-operative to 3-month post-activation interval | 1.4 [0.1 to 2.7]
  Speech: 3-month to 6-month post-activation interval | 0.7 [-0.1 to 1.5]
  Speech: 3-month to 9-month post-activation interval | 0.6 [-0.3 to 1.4]
  Speech: 3-month to 12-month post-activation interval | 0.7 [-0.1 to 1.6]
  Speech: 3-month to 18-month post-activation interval: number analyzed (Participants) | 19
  Speech: 3-month to 18-month post-activation interval | 0.8 [-0.0 to 1.6]
  Speech: 3-month to 24-month post-activation interval: number analyzed (Participants) | 19
  Speech: 3-month to 24-month post-activation interval | 0.9 [-0.1 to 1.9]
  Spatial: pre-operative to 3-month post-activation interval | 2.6 [0.9 to 4.2]
  Spatial: 3-month to 6-month post-activation interval | 0.8 [-0.4 to 1.9]
  Spatial: 3-month to 9-month post-activation interval | 1.0 [-0.3 to 2.3]
  Spatial: 3-month to 12-month post-activation interval | 1.3 [-0.1 to 2.6]
  Spatial: 3-month to 18-month post-activation interval: number analyzed (Participants) | 19
  Spatial: 3-month to 18-month post-activation interval | 1.7 [0.5 to 2.9]
  Spatial: 3-month to 24-month post-activation interval: number analyzed (Participants) | 19
  Spatial: 3-month to 24-month post-activation interval | 1.1 [-0.5 to 2.8]
  Qualities: pre-operative to 3-month post-activation interval | 1.0 [0.1 to 2.0]
  Qualities: 3-month to 6-month post-activation interval | 0.6 [-0.3 to 1.5]
  Qualities: 3-month to 9-month post-activation interval | 0.5 [-0.4 to 1.4]
  Qualities: 3-month to 12-month post-activation interval | 0.5 [-0.4 to 1.4]
  Qualities: 3-month to 18-month post-activation interval: number analyzed (Participants) | 19
  Qualities: 3-month to 18-month post-activation interval | 0.9 [0.0 to 1.9]
  Qualities: 3-month to 24-month post-activation interval: number analyzed (Participants) | 19
  Qualities: 3-month to 24-month post-activation interval | 0.4 [-0.5 to 1.4]
Statistical Analysis 1: Comparison: Cochlear Implant; Comparison of scores across time to investigate change in scores over time: Speech subtest; Test type: Superiority; p < 0.001, Mixed Models Analysis — The a priori threshold for statistical significance was p < 0.05
Statistical Analysis 2: Comparison: Cochlear Implant; Comparison of scores across time to investigate change in scores over time: Spatial subtest; Test type: Superiority; p = 0.001, Mixed Models Analysis — The a priori threshold for statistical significance was p < 0.05
Statistical Analysis 3: Comparison: Cochlear Implant; Comparison of scores across time to investigate change in scores over time: Qualities subtest; Test type: Superiority; p < 0.001, Mixed Models Analysis — The a priori threshold for statistical significance was p < 0.05

10. Primary Outcome: Change in Mean Response Scores as Measured by the Bern Single Sided Deafness (SSD) Questionnaire
Description: Bern SSD Questionnaire is a 10-item questionnaire used for rating perceived benefit of a hearing technology designed to be used for persons with Unilateral Hearing Loss (UHL). A positive score indicates greater perceived ability with the device and a negative score indicates greater perceived ability without the device. Scores range from -5 meaning much easier listening without the hearing device to +5 indicating much easier listening with the device. Scores across all 10 items are averaged for a single score. A modified version of this test that can be completed by a parent was used pre-operatively and at 3-, 6-, 9-, 12-, 18-, and 24-month post-activation intervals. Change is measured from the pre-operative to the 3-month post-activation interval and from the 3-month interval to each subsequent interval.
Time Frame: Pre-operatively through 24 months post-activation
Population: One participant was lost to follow-up after Month 12
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Cochlear Implant
Number analyzed (Participants) | 20
score on a scale
  Pre-operative to 3-month post-activation interval | 1.9 [0.8 to 3.0]
  3-month to the 6-month post-activation interval | 0.7 [0.0 to 1.4]
  3-month to the 9-month post-activation interval | 0.9 [0.2 to 1.6]
  3-month to the 12-month post-activation interval | 1.4 [0.7 to 2.1]
  3-month to the 18-month post-activation interval: number analyzed (Participants) | 19
  3-month to the 18-month post-activation interval | 1.5 [0.8 to 2.2]
  3-month to the 24-month post-activation interval: number analyzed (Participants) | 19
  3-month to the 24-month post-activation interval | 1.4 [0.7 to 2.1]
Statistical Analysis 1: Comparison: Cochlear Implant; Comparison of scores over time; Test type: Superiority; p < 0.001, Mixed Models Analysis — The a priori threshold for statistical significance was p < 0.05

11. Primary Outcome: Change in Mean Fatigue Scores as Measured by the Pediatric Quality of Life (PedsQL) Multidimensional Fatigue Scale
Description: PedsQL Multidimensional fatigue scale is a validated scale for determining fatigue in young children, including general fatigue, sleep/rest fatigue and cognitive fatigue. Scores from this test have been previously demonstrated to be substantially affected by hearing loss in children. A parent report version was used pre-operatively and at 3-, 6-, 9-, 12-, 18-, and 24-month post-activation intervals. Items are scored on a 5-point Likert scale and are then reversed scored and linearly transformed to a 0-100 scale where 100 would indicate no fatigue and 0 would indicate near constant fatigue.
Time Frame: Pre-operatively through 24 months post-activation
Population: One participant was lost to follow-up after Month 12
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Cochlear Implant
Number analyzed (Participants) | 20
score on a scale
  General Fatigue: pre-operative to 3-month post-activation | 5.4 [-4.2 to 15.1]
  General Fatigue: 3-month to 6-month post-activation | 4.6 [-5.1 to 14.2]
  General Fatigue: 3-month to 9-month post-activation | 1.9 [-7.8 to 11.5]
  General Fatigue: 3-month to 12-month post-activation | 2.5 [-71 to 12.2]
  General Fatigue: 3-month to 18-month post-activation: number analyzed (Participants) | 19
  General Fatigue: 3-month to 18-month post-activation | -1.0 [-10.8 to 8.8]
  General Fatigue: 3-month to 24-month post-activation: number analyzed (Participants) | 19
  General Fatigue: 3-month to 24-month post-activation | 4.0 [-5.8 to 13.8]
  Sleep Fatigue: Pre-operative to 3-month post-activation | 3.5 [-5.6 to 12.7]
  Sleep Fatigue: 3-month to 6-month post-activation | 6.5 [-2.6 to 15.6]
  Sleep Fatigue: 3-month to 9-month post-activation | 2.7 [-6.4 to 11.8]
  Sleep Fatigue: 3-month to 12-month post-activation | 2.7 [-6.4 to 11.8]
  Sleep Fatigue: 3-month to 18-month post-activation: number analyzed (Participants) | 19
  Sleep Fatigue: 3-month to 18-month post-activation | 4.2 [-5.1 to 13.4]
  Sleep Fatigue: 3-month to 24-month post-activation: number analyzed (Participants) | 19
  Sleep Fatigue: 3-month to 24-month post-activation | 3.5 [-5.7 to 12.8]
  Cognitive Fatigue: Pre-operative to 3-month post-activation | 7.5 [-3.4 to 18.4]
  Cognitive Fatigue: 3-month to 6-month post-activation | 3.3 [-7.5 to 14.2]
  Cognitive Fatigue: 3-month to 9-month post-activation | 0.8 [-10.0 to 11.7]
  Cognitive Fatigue: 3-month to 12-month post-activation | -2.3 [-13.2 to 8.6]
  Cognitive Fatigue: 3-month to 18-month post-activation: number analyzed (Participants) | 19
  Cognitive Fatigue: 3-month to 18-month post-activation | 1.7 [-9.3 to 12.8]
  Cognitive Fatigue: 3-month to 24-month post-activation: number analyzed (Participants) | 19
  Cognitive Fatigue: 3-month to 24-month post-activation | -2.2 [-13.2 to 8.8]
Statistical Analysis 1: Comparison: Cochlear Implant; Comparison of scores to evaluation change over time: General Fatigue Subtest; Test type: Superiority; p = 0.1009, Mixed Models Analysis — The a priori threshold for statistical significance was p < 0.05
Statistical Analysis 2: Comparison: Cochlear Implant; Comparison of scores to evaluation change over time: Sleep Fatigue Subtest; Test type: Superiority; p = 0.109, Mixed Models Analysis — The a priori threshold for statistical significance was p < 0.05
Statistical Analysis 3: Comparison: Cochlear Implant; Comparison of scores to evaluation change over time: Cognitive Fatigue Subtest; Test type: Superiority; p = 0.1733, Mixed Models Analysis — The a priori threshold for statistical significance was p < 0.05

ADVERSE EVENTS:
Time Frame: From the time of surgery through the Month 24 visit, a total of up to 25 months
Arm/Group | Cochlear Implant
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 4/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cochlear Implant (N=20)
Facial stimulation (Ear and labyrinth disorders) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Fall (General disorders) | 1 (1)
Sensory processing disorder (General disorders) | 1 (1)
Hearing loss progression in contralateral ear (Ear and labyrinth disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-13): https://cdn.clinicaltrials.gov/large-docs/74/NCT02963974/Prot_SAP_000.pdf